CLINICAL TRIAL: NCT00328367
Title: A Double-Blind Randomized Placebo Controlled Study of Aripiprazole Augmentation for Clozapine-Treated Patients With Refractory Schizophrenia
Brief Title: Aripiprazole Augmentation for Clozapine-Treated Patients With Refractory Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Yong Sik Kim/Professor, Seoul National University Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KYS-2006-05209
Record Dates: First submitted 2006-05-17; First posted 2006-05-19 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-04

CONDITIONS: Schizophrenia
Keywords: schizophrenia; aripiprazole; clozapine
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): clozapine plus aripiprazole
  Interventions: Drug: aripiprazole
- B (Placebo Comparator): clozapine plus placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: aripiprazole — aripiprazole augmentation of clozapine
  Other Names: abilify; OPC-14597
  Arms: A
Drug: placebo — placebo
  Arms: B

SUMMARY:
The purpose of this study is to determine whether aripiprazole augmentation is safe and effective in the treatment of clozapine-treated patients with refractory schizophrenia.

DETAILED DESCRIPTION:
Clozapine is renowned for its efficacy in treating schizophrenia refractory to typical or atypical antipsychotics. Though the effectiveness of clozapine has been established, a considerable number of patients with schizophrenia are partially responsive or unresponsive to clozapine. In addition, long-term use of clozapine is associated with the development of obsessive-compulsive symptoms and metabolic syndrome. In order to overcome these short-comings and to increase efficacy, aripiprazole augmentation was implemented. Quantitative electroencephalogram will be used to monitor the occurrence of abnormal findings and to analyze the changes in electroencephalographic pattern with linear and non-linear methodology.

Comparisons: Design of double-blind randomized placebo controlled study of patients at Refractory Schizophrenia Clinique in Department of Neuropsychiatry at Seoul National University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 18-65 years of age.
* Patients must have a diagnosis of schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV).
* Female patients of menarche must be using a medically accepted means of contraception (e.g. oral contraceptives, Depo-Provera, abstinence).
* Each patient must provide written informed consent after full explanation of study protocol, and authorized legal guardian must understand the nature of the study and must also give assent to study participation.
* Patients must have a baseline (day 0) BPRS score of at least 35 or over 2 of 5 SANS global rating item scores of at least 3.
* Patients have been receiving clozapine treatment for more than 1 year and there has been no change in clozapine dosage for more than 3 months.
* Patients must have a history of antipsychotic treatment with at least 2 different kinds prior to clozapine administration.
* Subjects who are fluent in Korean.

Exclusion Criteria:

* DSM-IV substance (except nicotine or caffeine) dependence within the past 1 year.
* Female patients who are either pregnant or lactating.
* Mental retardation (IQ < 70).
* Neurological disorders including epilepsy, stroke, or severe head trauma.
* Clinically significant laboratory abnormalities, on any of the following tests: CBC with differential, electrolytes, BUN, creatinine, hepatic transaminases, urinalysis and EKG.
* Prior history of aripiprazole non-response or intolerance.
* BPRS score of < 35 and over 4 of 5 SANS global rating item scores of < 3.
* Participation in a clinical trial of another investigational drug within 3 months (90 days) prior to study entry.
* Treatment with an injectable depot neuroleptic within less than three dosing interval between the last depot neuroleptic injections and baseline (day 0).
* History of electroconvulsive therapy within the past 3 months.
* Subjects who are not fluent in Korean.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2005-12; Primary Completion 2006-12 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Brief Psychotic Rating Scale (BPRS): Measure of efficacy will be changes in BPRS total and subscale scores from baseline to 8th week endpoint. Follow-up evaluation will be made every 6th month till 1 year after 8th week end point. | one year
Schedule for Assessment of Negative Symptoms (SANS): Measure of efficacy will be changes in SANS total and subscale scores from baseline to 8th week endpoint. Follow-up evaluation will be made at 6 month and 12 month after 8th week end point. | one year
Serum Prolactin Level | one year
Body Mass Index & Abdominal Circumference | one year
Lipid Panel with LDL Cholesterol | one year
FBS-PP & HbA1c | one year

SECONDARY OUTCOMES:
Clinical Global Impression-Severity & Improvement (CGI-S & CGI-I) | one year
Montgomery-Asberg Depression Rating Scale (MADRS) | one year
Yale-Brown Obsessive Compulsive Scale (YBOCS) | one year
Subjective Well-being under Neuroleptics scale (SWN) | one year
Drug-Induced Extrapyramidal Symptoms Scale (DIEPSS) | one year
Udvalg Fur Kliniske Undersogesler (UKU) | one year
Blood Pressure and Pulse Rate | one year
Admission Battery, CBC, & EKG | one year
Serum Clozapine Level | one year
Quantitative Electroencephalogram | one year

CONTACTS AND LOCATIONS:
Overall Officials: Yong Sik Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Rocha FL, Hara C. Benefits of combining aripiprazole to clozapine: three case reports. Prog Neuropsychopharmacol Biol Psychiatry. 2006 Aug 30;30(6):1167-9. doi: 10.1016/j.pnpbp.2006.03.024. Epub 2006 May 2. PMID 16647796
- [Background] Henderson DC, Kunkel L, Nguyen DD, Borba CP, Daley TB, Louie PM, Freudenreich O, Cather C, Evins AE, Goff DC. An exploratory open-label trial of aripiprazole as an adjuvant to clozapine therapy in chronic schizophrenia. Acta Psychiatr Scand. 2006 Feb;113(2):142-7. doi: 10.1111/j.1600-0447.2005.00612.x. PMID 16423166
- [Background] Ziegenbein M, Sieberer M, Calliess IT, Kropp S. Combination of clozapine and aripiprazole: a promising approach in treatment-resistant schizophrenia. Aust N Z J Psychiatry. 2005 Sep;39(9):840-1. doi: 10.1111/j.1440-1614.2005.01688_2.x. No abstract available. PMID 16168043
- [Derived] Chang JS, Ahn YM, Park HJ, Lee KY, Kim SH, Kang UG, Kim YS. Aripiprazole augmentation in clozapine-treated patients with refractory schizophrenia: an 8-week, randomized, double-blind, placebo-controlled trial. J Clin Psychiatry. 2008 May;69(5):720-31. doi: 10.4088/jcp.v69n0505. PMID 18370574
- See also: Click here for detailed information about aripiprazole. — http://www.nlm.nih.gov/medlineplus/druginfo/meds/a603012.html